CLINICAL TRIAL: NCT04964895
Title: Sexual Quality of Patients After Bladder Cancer Cystectomy : A Prospective Observational Study
Brief Title: Sexual Quality of Patients After Bladder Cancer Cystectomy
Acronym: QSCO
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/21/0113
Record Dates: First submitted 2021-07-06; First posted 2021-07-16 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2023-09

CONDITIONS: Sexual Dysfunction
Keywords: bladder cancer; cystectomy; sex life; sex quality
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Urinary Bladder Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with cystectomy
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Patients will fill in multiple questionnaires for this study :
  EORTC quality of life questionnaire (QLQ) QLQ-C30, EORTC Shq22, Male Sexual Health Questionnaire (MSHQ) only for Men, FSFI (only for women)

SUMMARY:
Bladder cancer is the second most prevalent urological cancer in France. About 1 in 5 new cases of bladder cancer infiltrate the muscles. The standard treatment is neoadjuvant chemotherapy followed by radical cystectomy associated with reconstruction of the urinary tract. The short-term effects on well-being and quality of life are well known. The long-term effects are, on the other hand, poorly understood, particularly sexual function. This study aim to asses the quality of sexual life in patients with cystectomy for bladder cancer. This will be done via various questionnaires given before and after surgery.

DETAILED DESCRIPTION:
The study is a prospective observational cohort study of the quality of sexual life in patients with cystectomy for bladder cancer. Data is collected via Qlq-C30, EORTC-Shq22, MSHQ if male, Female Sexual Function Index (FSFI) questionnaires that the patients complete by themselves. They are given before surgery and then 8 months after surgery.

The study consists of the compilation of relevant clinical data and questionnaire results.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient who had a cystectomy for bladder cancer
* Affiliated with a social security scheme

Exclusion Criteria:

* No Cystectomy
* Cystectomy for neurological etiology
* Pregnant or breastfeeding women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient who underwent cystectomy for bladder cancer during the study.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the decrease in the quality of sexual life of patients who had a cystectomy | T0 : before surgery
  EORTC SHQ C22 score before surgery
Evaluation of the decrease in the quality of sexual life of patients who had a cystectomy | T1 : 8 months after surgery
  EORTC SHQ C22 score 8 months after surgery

SECONDARY OUTCOMES:
Evaluation of the decrease in the quality of life of patients who had a cystectomy | T0 : before surgery
  QLQ-C30 score before surgery
Evaluation of the decrease in the quality of life of patients who had a cystectomy | T1 : 8 months after surgery
  QLQ-C30 score 8 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Eric Huyghe, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No